CLINICAL TRIAL: NCT05932056
Title: Miles de Manos (Thousands of Hands): Testing the Efficacy of a School-Based Youth Violence Preventive Intervention in a High Risk International Context
Brief Title: A Randomized Controlled Trial of Miles de Manos (Thousands of Hands)
Acronym: MdM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000446
Record Dates: First submitted 2023-06-15; First posted 2023-07-06 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Miles de Manos (Thousands of Hands) Intervention (Experimental): Parents and teachers from schools randomized to this arm will receive the Miles de Manos (Thousands of Hands) intervention. Miles de Manos (Thousands of Hands) comprises 3 components: a cognitive-behavioral skills training component for parents (8 sessions), a cognitive-behavioral skills training component for school staff (10 sessions), and a "bridge" component that brings parents, teachers, and school administrators together to talk about how to support each other's efforts related to youth violence prevention (4 sessions). Core elements include effective communication, clear expectations, limits and consequences, positive reinforcement, adult supervision and monitoring, effective problem solving, and emotion regulation. Miles de Manos (Thousands of Hands) is highly interactive and involves brief lectures, small and large group discussions, role-plays, and interactive exercises.
  Interventions: Behavioral: Miles de Manos (Thousands of Hands)
- Control (No Intervention): Parents and teachers from schools randomized to this arm will receive services as usual as provided by their schools.

INTERVENTIONS:
Behavioral: Miles de Manos (Thousands of Hands) — Miles de Manos (Thousands of Hands) is a school-based group intervention that incorporates elements of evidence-based behavior management interventions in parent, teacher, and parent-teacher joint sessions.
  Arms: Miles de Manos (Thousands of Hands) Intervention

SUMMARY:
Violence is one of the leading causes of death for young people and has widespread costs for individuals, families and communities. This study will test the effectiveness of Miles de Manos (Thousands of Hands), a group-based violence prevention program for elementary school students in Honduras. Miles de Manos (Thousands of Hands) has three components: parents/caregiver groups, teacher groups, and groups that combine parents/caregivers and teachers together. The study will examine the program's impact on parent and teacher's behaviors as well as student behavior problems.

DETAILED DESCRIPTION:
The purpose of this study, a randomized controlled trial, is to examine the outcomes, and potential mediators and moderators of those outcomes, related to a school-based youth violence program, Miles de Manos (Thousands of Hands; MdM), delivered within public primary schools within the country of Honduras. Miles de Manos (Thousands of Hands), which is conducted with parents/caregivers and teachers, was developed through a collaboration of a multinational group of practitioners, educators, administrators, scientists, and curriculum writers from Honduras, El Salvador, Guatemala, Nicaragua, Germany, and the United States with funding from the German non-governmental organization Deutsche Gesellschaft für Internationale Zusammenarbeit (GIZ). It is similar in core content to evidence-based programs that were developed in the United States. During the development process, the program was piloted tested in Honduras multiple times, and is currently being employed in public primary schools across Honduras. The aims of the study are as follows:

Aim 1. To examine the effectiveness of a culturally specified youth violence prevention program on improving effective parent and teacher behavior management practices and reducing both youth problem behaviors and youth association with peers and adults involved in problem behaviors.

Aim 2. To investigate potential mediators of any outcomes due to the intervention, and specifically to conduct a test of the social learning theory underlying the intervention.

Aim 3. To investigate potential moderators of any outcomes due to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Students in grades 3-5, and their parents and teachers, from participating schools located in neighborhoods in and around Tegucigalpa, Honduras.
* Inclusion criteria for participating schools will include those with no prior implementation of Miles de Manos (Thousands of Hands); school location will be in urban or semi-urban areas; and adequate school engagement and commitment from staff and school leaders, parents, community leaders, and community institutions and officials.

Exclusion Criteria:

* Schools with prior implementation of Miles de Manos (Thousands of Hands) will not be eligible to participate.

Ages: 7 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Child conduct problems (baseline) | Child conduct problems are measured at baseline.
  Child conduct problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Child conduct problems (6-9 months) | Child conduct problems are measured at 6-9 months post-baseline after the termination of the Miles de Manos (Thousands of Hands) program in intervention schools.
  Child conduct problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Child conduct problems (12-15 months) | Child conduct problems are measured at about 1 year post-baseline
  Child conduct problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Change from baseline child conduct problems to 6-9 months | Change in child conduct problems between baseline and 6-9 months.
  Child conduct problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Change from baseline child conduct problems to about 1 year post-baseline | Change in child conduct problems between baseline and about 1 year post-baseline.
  Child conduct problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Child hyperactivity/inattention (baseline) | Child hyperactivity/inattention is measured at baseline.
  Child hyperactivity/inattention is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Child hyperactivity/inattention (6-9 months) | Child hyperactivity/inattention is measured at 6-9 months post-baseline after the termination of the Miles de Manos (Thousands of Hands) program in intervention schools.
  Child hyperactivity/inattention is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Child hyperactivity/inattention (12-15 months) | Child hyperactivity/inattention is measured at about 1 year post-baseline.
  Child hyperactivity/inattention is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Change from baseline child hyperactivity/inattention to 6-9 months | Change in baseline child hyperactivity/inattention to 6-9 months.
  Child hyperactivity/inattention is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Change from baseline child hyperactivity/inattention to about 1 year | Change from baseline child hyperactivity/inattention to about 1 year post-baseline
  Child hyperactivity/inattention is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Child emotional problems (baseline) | Child emotional problems are measured at baseline.
  Child emotional problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Child emotional problems (6-9 months) | Child emotional problems are measured at 6-9 months post-baseline after the termination of the Miles de Manos (Thousands of Hands) program in intervention schools..
  Child emotional problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Child emotional problems (12-15 months) | Child emotional problems are measured at about 1 year post-baseline.
  Child emotional problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Change in baseline child emotional problems to 6-9 months | Change in baseline child emotional problems to 6-9 months
  Child emotional problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Change in baseline child emotional problems to about 1 year | Child emotional problems are measured at about 1 year post-baseline.
  Child emotional problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Child peer relationship problems (baseline) | Child peer relationship problems are measured at baseline.
  Child peer relationship problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Child peer relationship problems (6-9 months) | Child peer relationship problems are measured at 6-9 months post-baseline after the termination of the Miles de Manos (Thousands of Hands) program in intervention schools.
  Child peer relationship problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Child peer relationship problems (12-15 months) | Child peer relationship problems are measured at about 1 year post-baseline.
  Child peer relationship problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Change in baseline child peer relationship problems to 6-9 months | Change in baseline child peer relationship problems to 6-9 months
  Child peer relationship problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Change in baseline child peer relationship problems to about 1 year | Change in baseline child peer relationship problems to about 1 year
  Child peer relationship problems is a sub-scale of the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire about 2-17 year olds. The SDQ response scale consists of 3 choices: 0-not true; 1-somewhat true; 2-certainly true. The sub-scale for conduct problems includes the mean score of 5 items.
Parenting (baseline) | Parenting is measured at baseline.
  The parenting outcome is a sub-scale of the Parent and Family Adjustment Scales (PAFAS). The PAFAS was designed as a brief outcome measure for assessing changes in parenting practices in the evaluation of group parenting interventions. The inventory consists of the Parenting scale measuring parenting practices and quality of parent-child relationship and of the Family Adjustment scale measuring parental emotional adjustment and partner and family support in parenting. All items are scored from 0 to 3 with the parenting sub-scale reflecting a sum score of 4 sub-scales totaling 21 items that focus on: parental consistency, coercive parenting, positive encouragement, and parent-child relationship.
Parenting (6-9 months) | Parenting is measured at 6-9 months post-baseline after the termination of the Miles de Manos (Thousands of Hands) program in intervention schools.
  The parenting outcome is a sub-scale of the Parent and Family Adjustment Scales (PAFAS). The PAFAS was designed as a brief outcome measure for assessing changes in parenting practices in the evaluation of group parenting interventions. The inventory consists of the Parenting scale measuring parenting practices and quality of parent-child relationship and of the Family Adjustment scale measuring parental emotional adjustment and partner and family support in parenting. All items are scored from 0 to 3 with the parenting sub-scale reflecting a sum score of 4 sub-scales totaling 21 items that focus on: parental consistency, coercive parenting, positive encouragement, and parent-child relationship.
Parenting (12-15 months) | Parenting is measured at about 1 year post-baseline.
  The parenting outcome is a sub-scale of the Parent and Family Adjustment Scales (PAFAS). The PAFAS was designed as a brief outcome measure for assessing changes in parenting practices in the evaluation of group parenting interventions. The inventory consists of the Parenting scale measuring parenting practices and quality of parent-child relationship and of the Family Adjustment scale measuring parental emotional adjustment and partner and family support in parenting. All items are scored from 0 to 3 with the parenting sub-scale reflecting a sum score of 4 sub-scales totaling 21 items that focus on: parental consistency, coercive parenting, positive encouragement, and parent-child relationship.
Change in baseline parenting to 6-9 months. | Change in baseline parenting to 6-9 months.
  The parenting outcome is a sub-scale of the Parent and Family Adjustment Scales (PAFAS). The PAFAS was designed as a brief outcome measure for assessing changes in parenting practices in the evaluation of group parenting interventions. The inventory consists of the Parenting scale measuring parenting practices and quality of parent-child relationship and of the Family Adjustment scale measuring parental emotional adjustment and partner and family support in parenting. All items are scored from 0 to 3 with the parenting sub-scale reflecting a sum score of 4 sub-scales totaling 21 items that focus on: parental consistency, coercive parenting, positive encouragement, and parent-child relationship.
Change in baseline parenting to about 1 year. | Change in baseline parenting to about 1 year.
  The parenting outcome is a sub-scale of the Parent and Family Adjustment Scales (PAFAS). The PAFAS was designed as a brief outcome measure for assessing changes in parenting practices in the evaluation of group parenting interventions. The inventory consists of the Parenting scale measuring parenting practices and quality of parent-child relationship and of the Family Adjustment scale measuring parental emotional adjustment and partner and family support in parenting. All items are scored from 0 to 3 with the parenting sub-scale reflecting a sum score of 4 sub-scales totaling 21 items that focus on: parental consistency, coercive parenting, positive encouragement, and parent-child relationship.
Family adjustment (baseline) | Family adjustment is measured at baseline.
  The family adjustment outcome is a sub-scale of the Parent and Family Adjustment Scales (PAFAS). The PAFAS was designed as a brief outcome measure for assessing changes in parental adjustment in the evaluation of group parenting interventions. The inventory consists of the Parenting scale measuring parenting practices and quality of parent-child relationship and of the Family Adjustment scale measuring parental emotional adjustment and partner and family support in parenting. All items are scored from 0 to 3 with the parenting sub-scale reflecting a sum score of 3 sub-scales totaling 9 items that focus on: parental adjustment, family relationships, and parental teamwork.
Family adjustment (6-9 months) | Family adjustment is 6-9 months post-baseline after the termination of the Miles de Manos (Thousands of Hands) program in intervention schools.
  The family adjustment outcome is a sub-scale of the Parent and Family Adjustment Scales (PAFAS). The PAFAS was designed as a brief outcome measure for assessing changes in parental adjustment in the evaluation of group parenting interventions. The inventory consists of the Parenting scale measuring parenting practices and quality of parent-child relationship and of the Family Adjustment scale measuring parental emotional adjustment and partner and family support in parenting. All items are scored from 0 to 3 with the parenting sub-scale reflecting a sum score of 3 sub-scales totaling 9 items that focus on: parental adjustment, family relationships, and parental teamwork.
Family adjustment (12-15 months) | Family adjustment is measured at about 1 year post-baseline.
  The family adjustment outcome is a sub-scale of the Parent and Family Adjustment Scales (PAFAS). The PAFAS was designed as a brief outcome measure for assessing changes in parental adjustment in the evaluation of group parenting interventions. The inventory consists of the Parenting scale measuring parenting practices and quality of parent-child relationship and of the Family Adjustment scale measuring parental emotional adjustment and partner and family support in parenting. All items are scored from 0 to 3 with the parenting sub-scale reflecting a sum score of 3 sub-scales totaling 9 items that focus on: parental adjustment, family relationships, and parental teamwork.
Change in baseline family adjustment to 6-9 months | Change in baseline family adjustment to 6-9 months
  The family adjustment outcome is a sub-scale of the Parent and Family Adjustment Scales (PAFAS). The PAFAS was designed as a brief outcome measure for assessing changes in parental adjustment in the evaluation of group parenting interventions. The inventory consists of the Parenting scale measuring parenting practices and quality of parent-child relationship and of the Family Adjustment scale measuring parental emotional adjustment and partner and family support in parenting. All items are scored from 0 to 3 with the parenting sub-scale reflecting a sum score of 3 sub-scales totaling 9 items that focus on: parental adjustment, family relationships, and parental teamwork.
Change in baseline family adjustment to about 1 year | Change in baseline family adjustment to about 1 year
  The family adjustment outcome is a sub-scale of the Parent and Family Adjustment Scales (PAFAS). The PAFAS was designed as a brief outcome measure for assessing changes in parental adjustment in the evaluation of group parenting interventions. The inventory consists of the Parenting scale measuring parenting practices and quality of parent-child relationship and of the Family Adjustment scale measuring parental emotional adjustment and partner and family support in parenting. All items are scored from 0 to 3 with the parenting sub-scale reflecting a sum score of 3 sub-scales totaling 9 items that focus on: parental adjustment, family relationships, and parental teamwork.
Teacher classroom behavior management (baseline) | Teacher classroom behavior management is measured at baseline.
  This outcome is measured using the Positive Behavior Intervention and Supports (PBIS) Positive Behavior Support Classroom Management: Self-Assessment Revised. This brief 10-item survey is focused on teacher classroom strategies to support the prosocial behaviors and high academic and social engagement of their students.
Teacher classroom behavior management (6-9 months) | Teacher classroom behavior management is measured at 6-9 months post-baseline after the termination of the Miles de Manos (Thousands of Hands) program in intervention schools.
  This outcome is measured using the Positive Behavior Intervention and Supports (PBIS) Positive Behavior Support Classroom Management: Self-Assessment Revised. This brief 10-item survey is focused on teacher classroom strategies to support the prosocial behaviors and high academic and social engagement of their students.
Teacher classroom behavior management (12-15 months) | Teacher classroom behavior management is measured at about 1 year post-baseline.
  This outcome is measured using the Positive Behavior Intervention and Supports (PBIS) Positive Behavior Support Classroom Management: Self-Assessment Revised. This brief 10-item survey is focused on teacher classroom strategies to support the prosocial behaviors and high academic and social engagement of their students.
Change in baseline teacher classroom behavior management to 6-9 months | Change in baseline teacher classroom behavior management to 6-9 months
  This outcome is measured using the Positive Behavior Intervention and Supports (PBIS) Positive Behavior Support Classroom Management: Self-Assessment Revised. This brief 10-item survey is focused on teacher classroom strategies to support the prosocial behaviors and high academic and social engagement of their students.
Change in baseline teacher classroom behavior management to about 1 year | Change in baseline teacher classroom behavior management to about 1 year
  This outcome is measured using the Positive Behavior Intervention and Supports (PBIS) Positive Behavior Support Classroom Management: Self-Assessment Revised. This brief 10-item survey is focused on teacher classroom strategies to support the prosocial behaviors and high academic and social engagement of their students.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make personally deidentified data sets available to other researchers that include individual data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After 7/31/2024 when we complete analyses for our primary endpoint.
Access Criteria: Data will be provided upon request.